CLINICAL TRIAL: NCT02104908
Title: Target-controlled Propofol Infusion as a Technique of Anesthesia for Surgery of Hip Fracture Under Ultrasound Guidance Lumbar and Sacral Plexus Block or Lumbar, Sacral and Paravertebral Nerve Block in the Elderly
Brief Title: Study of Nerve Block Anesthesia for Surgery of Hip Fracture in the Elderly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Daqiang Zhao, Daqiang Zhao, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARA-2014
Record Dates: First submitted 2014-03-03; First posted 2014-04-07 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-01

CONDITIONS: Anesthesia; Reaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paravertebral nerve (Experimental): Injection with 20ml 0.5% ropivacaine at lumbar plexus(level L3-4) , 10ml 0.5%ropivacaine at sacral plexus and 10ml 0.5%ropivacaine at paravertebral nerve(level L1)
  Interventions: Procedure: paravertebral nerve
- lumbar and sacral plexus block (Other): a lumbar and sacral plexus block(LS) group with 20ml 0.5% ropivacaine at lumbar plexus(level L3-4) and 10ml 0.5%ropivacaine at sacral plexus;
  Interventions: Procedure: lumbar and sacral plexus block

INTERVENTIONS:
Procedure: paravertebral nerve — a lumbar, sacral plexus and paravertebral nerve block(LSP) group with 20ml 0.5% ropivacaine at lumbar plexus(level L3-4) , 10ml 0.5%ropivacaine at sacral plexus and 10ml 0.5%ropivacaine at paravertebral nerve(level L1).
  Arms: paravertebral nerve
Procedure: lumbar and sacral plexus block — a lumbar and sacral plexus block(LS) group with 20ml 0.5% ropivacaine at lumbar plexus(level L3-4) and 10ml 0.5%ropivacaine at sacral plexus;
  Arms: lumbar and sacral plexus block

SUMMARY:
The investigators aim to examine target-controlled propofol infusion as a technique of anesthesia for surgery of hip fracture under ultrasound guidance lumbar and sacral plexus block or lumbar, sacral and paravertebral nerve block in the elderly; and to evaluate which regional anesthesia was more sufficient for the old.

DETAILED DESCRIPTION:
Eighty patients with American Society of Anesthesiologists（ASA） Ⅰ-Ⅲ older than 80 years are randomly assigned to 2 groups: a lumbar and sacral plexus block(LS) group with 20ml 0.5% ropivacaine at lumbar plexus(level L3-4) and 10ml 0.5%ropivacaine at sacral plexus; a lumbar, sacral plexus and paravertebral nerve block(LSP) group with 20ml 0.5% ropivacaine at lumbar plexus(level L3-4) , 10ml 0.5%ropivacaine at sacral plexus and 10ml 0.5%ropivacaine at paravertebral nerve(level L1). The target-controlled propofol infusion is started immediately after positioning the patient on the operating table. The initial target concentration was 0.5μg/mL. The infusion rate is adjusted every 5min by increasing or decreasing the target concentration by 0.2μg/mL steps based on the patients' respiratory rate(RR), blood pressure(BP), heart rate(HR), and level of sedation(score of 5 on Ramsay Sedation Scale ). The minimal, maximal, optimal target concentration, cumulative propofol dose, frequency of spontaneous movement and incidences of associated complications are recorded. Patients were phoned for followup and questioned for activity status in one year. If the patients were dead, date of death; if they survived, daily living activity questioned.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ-Ⅲ
* hip fracture need surgery

Exclusion Criteria:

* patient refusal
* chronic use of opioids
* coagulation disorders
* preexisting neurological disorders

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
cumulative propofol dose | 24 weeks

SECONDARY OUTCOMES:
The optimal target concentration propofol | 24 weeks

OTHER OUTCOMES:
Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daqiang Zhao, Master, Principal Investigator — Shanghai Jiaotong University Affiliated Sixth People's Hospital Shanghai,China